CLINICAL TRIAL: NCT03891277
Title: Efficacy and Safety of Ferrous Iron on the Prevention of Vascular Cognitive Impairment Among Patients With Cerebral Infarction/TIA,FAVORITE
Brief Title: Efficacy and Safety of Ferrous Iron on the Prevention of Vascular Cognitive Impairment Among Patients With Cerebral Infarction/TIA (FAVORITE)
Acronym: FAVORITE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, 86(010)59978351, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018YFC1312303
Record Dates: First submitted 2019-02-25; First posted 2019-03-27 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Vascular Cognitive Impairment; Dementia, Vascular; Iron-deficiency; Cerebral Infarction; TIA
Keywords: Vascular Cognitive Impairment; dementia; iron deficiency; cerebral infarction; TIA; biological markers; Clinical Trial
MeSH Terms: conditions — Dementia, Vascular; Anemia, Iron-Deficiency; Cerebral Infarction; Dementia; Iron Deficiencies | interventions — ferrous succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two nearly identical tablet forms of Ferrous iron (0.2g Ferrous iron and matching placebo) with almost the same size, color and smell will be used in this research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferrous succinate (Active Comparator): Ferrous succinate sustained-release tablets（Ferrous succinate 0.2g）1 tablet, Qd, po during or after breakfast, Lasting for 12 weeks.
  Interventions: Drug: Ferrous succinate
- placebo (Placebo Comparator): placebo with almost the same size, color and smell as Ferrous iron will be used with 1 tablet, Qd, po during or after breakfast, Lasting for 12 weeks.
  Interventions: Drug: Ferrous succinate

INTERVENTIONS:
Drug: Ferrous succinate — Ferrous succinate sustained-release tablets（Ferrous succinate 0.2g）1 tablet, Qd,po during or after breakfast, Lasting for 12 weeks.
  placebo with almost the same size, color and smell as Ferrous iron will be used with 1 tablet, Qd, po during or after breakfast, Lasting for 12 weeks.
  Other Names: Placebo

SUMMARY:
The prevalence of Vascular Cognitive Impairment(VCI) is high in patients after ischemic stroke or transient ischemic attack(TIA) . Effective therapy for the prevention of VCI remains limited. The primary purpose of this study is to evaluate the efficacy and safety of Ferrous iron versus placebo on the prevention of vascular cognitive impairment among patients with ischemic stroke/TIA complicated with Hemoglobin deficiency.

DETAILED DESCRIPTION:
The prevalence of Vascular Cognitive Impairment(VCI) remains 21%~70% among patients after ischemic stroke or TIA. Effective therapy for the prevention of VCI remains limited. Abnormal iron distribution and Systemic iron deficiency may contribute partly to the occurrence of VCI.The primary purpose of this study is to evaluate the efficacy and safety of Ferrous iron versus placebo in reducing the risk of VCI at 1 year in patients with cerebral Infarction/TIA complicated with Hemoglobin deficiency. The secondary purpose is to evaluate the effect of Ferrous iron on the Biological markers of VCI; to evaluate the effect of iron supplement on the outcome(death,stroke recurrence, dependency) of patients with ischemic stroke or TIA complicated with Hemoglobin deficiency at 3 months/1 year after treatment.

This trial is a randomized, double-blind, placebo-controlled, multicenter clinical trial. 1006 patients in 20 centers in China will be enrolled with one of the following situations 1.recent ischemic stroke or TIA (within 3 months) with Fe deficiency （serum ferritin<20µg/L）or Hemoglobin deficiency(<120g/L for female and <130g/L for male).2. Vascular risk factors(hypertension, diabetes mellitus, or dyslipidemia), with multiply lacunar infarctions(≥2) or extensive white matter lesions（Fazekas ≥2） or multiply microhaemorrhage(≥2) showed on CT/Magnetic Resonance(MR) with Fe deficiency （serum ferritin<20µg/L）or Hemoglobin deficiency(<120g/L for female and <130g/L for male).. Patients will be randomly assigned into 2 groups according to the ratio of 1:1:

Ferrous iron therapy (0.2 per day) Placebo Face to face interviews will be made at baseline, 14 (or hospital discharge), 3th month± 7 days and 12th month ± 14 days after randomization.

Primary outcome is defined as prevalence of Vascular Cognition Impairment at 1 year after treatment. Secondary outcomes include all-cause death; ischemic stroke; transient ischemic attack; poor functional outcome (mRS 2-6). Safety outcomes, relating to adverse gastrointestinal reactions and iron overload.

ELIGIBILITY:
Inclusion Criteria:

1. Age :18-80 years old , male or female;
2. one of the following situations: A.recent ischemic stroke or TIA (within 3 months) B. One or more vascular risk factors including hypertension, diabetes mellitus, or dyslipidemia, with multiply lacunar infarctions(≥2) or extensive white matter lesions（Fazekas ≥2） or multiply microhaemorrhage(≥2) showed on CT/MR.
3. Fe deficiency （serum ferritin<20µg/L）or Hemoglobin deficiency(≥60 g/L and <120g/L for female,or ≥60 g/L and <130g/L for male)
4. Signed informed consent.

Exclusion Criteria:

1. CT/MR showed Intracranial haemorrhage or non-cerebral vascular disease (eg. intracranial tumors, multiple sclerosis);
2. Patients who Can not cooperate with the completion of neuropsychological evaluation for Severe hearing impairment, visual impairment, unilateral neglect, or dyskinesia;
3. Patients with Severe anemia with Hemoglobin<60 g/L;
4. Patients with thalassemia, megaloblastic anemia or erythronoclastic anemia.
5. Patients with Mental illness or schizophrenia;
6. Patients who were diagnosed definitely as Alzheimer's disease;
7. Patients having history of taking drugs including Cholinesterase inhibitors、NMDA antagonists、5-hydroxytryptophan receptor antagonists、pyrrolidone and other definite drugs for improving cognition(e.g. donepezil、Galanthamine、Memantine、huperzine A、oxiracetam、aniracetam、piracetam、butyphthalide) within 3 months before randomization；
8. Patients with severe liver or kidney insufficiency(ALT>twofold upper normal limit or Aspartate Aminotransferase>twofold upper normal limit; Cr>1.5 times upper normal limit or Glomerular Filtration Rate<40 ml/min/1.73m2）;
9. Patients with Severe untreated urinary tract infection;
10. Patients with hemochromatosis or hemosiderosis(e.g. Iron lung deposition);
11. Patients with Iron allergy or other contraindications of using Iron；
12. Pregnant or childbearing-age women；
13. Patients who are undergoing experimental drugs or device tests;
14. Patients Unable to finish the follow-up of 3 months or 1 year due to geographical factor or other reasons;
15. Patients or legal representatives refuse to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of vascular cognitive impairment in patients given Ferrous succinate versus placebo | 1 year after randomization
  Vascular cognitive impairment will be diagnosed with Montreal Cognitive Assessment(MoCA, range 0-30 scores) <26 scores

SECONDARY OUTCOMES:
All-cause death | 1 year after randomization
  All-cause death
Stroke recurrence (including hemorrhagic and ischemic stroke) | 1 year after randomization
  Stroke recurrence including hemorrhagic and ischemic stroke
Poor functional outcome | 1 year after randomization
  The modified Rankin Scale (mRS range 0-6)= 2-6
Value of Hemoglobin/serum ferritin/serum Tau/serum Aß | 3 months and 1 year after randomization
  Value of Hemoglobin/serum ferritin/serum Tau/serum Aß

CONTACTS AND LOCATIONS:
Overall Officials: Jia Qian, doctor, Study Chair — Beijing Tiantan Hospital; Zhang shuting, doctor, Study Director — West China Hospital
Locations (1):
- Beijing tiantan hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jia Q, Lei P, Sun L, Jia WL, Pan Y, Yuan B, Wang Y, Zhou Q, Meng X, Jing J, Lin J, Wang A, Zhang S, Hong Z, Yang Y, Xiong Y, Li Z, Wang Y, Zhao X, Wang Y. Efficacy and safety of Ferrous iron on the prevention of Vascular cOgnitive impaiRment among patients with cerebral Infarction/TIA (FAVORITE): rationale and design of a multicentre randomised trial. Stroke Vasc Neurol. 2025 Feb 25;10(1):136-141. doi: 10.1136/svn-2023-002644. PMID 38789134